CLINICAL TRIAL: NCT02063815
Title: A Randomized Controlled Trial of Caries Prevention Effect of a Glass Ionomer Sealant Versus a Resin Sealant
Brief Title: A Trial of Caries Prevention Effect of Fissure Sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAG-A-040609-0167
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Caries Prevention; Fissure Sealant; Fluoride Concentration; Glass Ionomer Cement; Resin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- glass ionomer based fissure sealant (Active Comparator): fissure sealant application
  Interventions: Procedure: Fissure sealant application
- resin based fissure sealant (Active Comparator): fissure sealant application
  Interventions: Procedure: Fissure sealant application

INTERVENTIONS:
Procedure: Fissure sealant application

SUMMARY:
The purpose of this randomized clinical trial was to compare caries prevention of a conventional resin-based sealant and a glass-ionomer sealant placed on occlusal pits and fissures over a one year period in a high caries children group. Additionally the concentration of Fluoride in saliva was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age range of 6 to 10 years 2.Having caries free, fully erupted first permanent molars 3.Deep and/or intermediate pits or fissures 4.dft ≥ 2

Exclusion Criteria:

* 1.Having any systemic disease 2.Topical fluoride was applied last six months 3.dft = 0

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Fluoride concentration of saliva | 1 week, 6. months, 12. months